CLINICAL TRIAL: NCT06042283
Title: Assessing the Efficacy of Metacognitive Training on Depressive Symptoms, Dysfunctional Attitudes and Metacognition in Older Adults Diagnosed With Depression
Brief Title: Efficacy of Metacognitive Training in Older Adults With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Lect. Merve MURAT MEHMED ALİ, Ph.D.(c), MSN, RN, Lecturer & Ph.D. Student at Psychiatric Mental Health Nursing Department, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 01
Record Dates: First submitted 2023-08-15; First posted 2023-09-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Depression in Old Age
Keywords: geriatric depression; psychotherapy; metacognitive training-silver; thought distortions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will have Metacognitive Training-Silver program. Metacognitive Training-Silver program is an eight-module training that focuses on common cognitive problems and dysfunctional attitudes, beliefs and prejudices in solving problems seen in depression. The purpose of the sessions is to convey information about false beliefs and cognitive distortions, and to help sick individuals think critically, convey their thoughts, and acquire new problem-solving strategies through exercises.
  Interventions: Behavioral: Metacognitive Training-Silver
- Control group (No Intervention): All participants in the control group will continue the treatment process determined in the routine. In this process, the patient participates in counseling and/or psychotherapy, ECT (electroconvulsive therapy) sessions, and psychopharmacological drugs. The control group will not participate in the Metacognitive Training-Silver program, an interview consisting of one session is planned considering for the placebo effect. At the end of the study, the Metacognitive Training-Silver program will be carried out with the voluntary participants in the control group, taking into account the ethics.

INTERVENTIONS:
Behavioral: Metacognitive Training-Silver — The Metacognitive Training-Silver program includes the following topics: Thinking and Reasoning 1 (module 1), Memory (module 2), Thinking and Reasoning 2 (module 3), Self-Esteem (module 4), Thinking and Reasoning 3 (module 5), Behaviors and Strategies (module 6), Thinking and Reasoning 4 (module 7) and Perception of Feelings (module 8).
  Each session is planned to last 45-60 minutes. Materials will be used in the Metacognitive Training-Silver program are PPT (Power Point Presentations) slides, videos, homework exercises, and yellow-red cards.
  Metacognitive Training-Silver is planned to be applied face-to-face in 3 groups (12, 10, and 10 people) at scheduled times in a quiet room suitable for the group. In order to increase compliance with the Metacognitive Training-Silver program, the sessions will be applied during the routine treatment period.
  Arms: Intervention Group

SUMMARY:
Effective pharmacological and psychological treatments for depression are available. However, treatment modalities are not accessible to all patients diagnosed with depression. Furthermore, some individuals who access treatment drop out and relapse after treatment. Improving treatment modalities for depression is important given the rates of individuals diagnosed worldwide, and rather than developing new treatments, there is a need to explore how existing treatment modalities can be improved and implemented in a simpler and more cost-effective way. To address this need, Metacognitive Training for Depression (DMCT) was developed as a low-cost, easy-to-implement, cognitive behavioral therapy-based group intervention. The aim of Metacognitive Training is to reduce depressive symptoms by working with the patient's cognitive biases from a metacognitive perspective. The effectiveness of this method, which has been proven effective by studies in the literature, is presented with a pilot study on older adults in 2018. Since the studies evaluating the effectiveness of the Metacognitive Training-Silver program are limited and it has not yet been adapted to Turkish culture, this study aims to evaluate the effectiveness of the Metacognitive Training-Silver program in older adults diagnosed with depression.

DETAILED DESCRIPTION:
According to the Global Burden of Disease (GBD-2019) report, mental disorders have been at the top of the global burden of disease list between 1990 and 2019. Depression ranks first among mental disorders with disability and psychosocial dependence. The worldwide prevalence rate of depression is 3.8% and it is a common disorder. The prevalence rate in adults is 5%, and the prevalence rate in adults aged 60 and over is 5.7%. According to the 2021 data from the US Centers for Disease Control and Prevention, compared to the general population, the rate of depression is 13.5% higher in older adults who need home healthcare services and 11.5% higher in hospitalized older adults. A recent systematic review and meta-analysis (2022) found that the global prevalence rate of depression in older adults was 28.4% and that the prevalence of depression in older adults is high, although there are variations by geographical location, diagnostic/screening tools, sample size, representativeness, and study quality. The isolation measures taken to prevent the spread of the COVID-19 pandemic have negative psychological effects on the protection of vulnerable groups, including older adults. Therefore, the pandemic is reported to have led to a significant increase in major depression cases globally, with an estimated 28.1% increase. With the COVID-19 pandemic, there is an increase in the demand for mental health services due to the increase in the incidence of depression and anxiety. Depression is more than a short-term emotional response to mood swings and psychological difficulties experienced in daily life. Especially recurrent and moderate or severe depression is an important health problem. The individual's daily life is negatively affected, functionality decreases and/or suicide may occur.

Depression is a serious mental disorder characterized by symptoms such as depressed mood or loss of interest/desire. In addition to these important symptoms, DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) criteria include sleep problems, changes in appetite/weight, psychomotor restlessness/agitation, loss of energy, concentration problems, feelings of worthlessness or guilt, and recurrent suicidal thoughts. Over time, this illness leads to cognitive and social dysfunction.

In the treatment of depression, multimodal treatment options need to be carried out simultaneously. Although there are known effective treatments for mental disorders, more than 75% of people in low- and middle-income countries do not receive treatment. Barriers to effective care include a lack of financial resources, lack of legal regulations, lack of trained health professionals, and stigma. Therefore, psychotherapeutic interventions in inpatient/outpatient mental health facilities for psychosocial rehabilitation are insufficient, and effective care management is needed to address this problem.

In the treatment of depression, only medication can be used due to various factors such as patient preference and economic reasons. However, despite medication, the disability and decreased functionality seen in patients are not sufficient for the rehabilitation of the patient. Insight into the disease and low compliance with treatment emphasizes the need for psychotherapies and psychosocial interventions. In this sense, cognitive-behavioral therapy approaches and family interventions are an essential complement to psychopharmacology.

Metacognitive Training (MCT) was created by Steffen Moritz (2007) focusing on psychosis. Studies conducted using MCT show that MCT is beneficial in patients with schizophrenia and psychosis, reduces the severity of delusions, and shows a positive effect even after 6 months of follow-up. Following these results, Metacognitive Training for Depression (D-MCT), which focuses on cognitive biases specific to depression, was developed based on the Metacognitive Training for Psychosis program. Metacognitive Training for Depression is a new treatment option for depression and is a variant of cognitive behavioral therapy that adopts a metacognitive perspective by focusing on changing cognitive biases and dysfunctional attitudes. In the first pilot study conducted by Jelinek et al. (2013), it was proven that there was a significant decrease in depressive symptoms, cognitive distortions, and rumination and an increase in self-esteem. In other randomized controlled studies conducted by Jelinek and colleagues, at the end of Metacognitive Training for Depression and at 6-month follow-up, it was determined that there was more improvement in depressive symptoms and a decrease in dysfunctional metacognitive beliefs. In secondary analyses conducted 3.5 years later, it was found that positive effects were still seen in the groups where Metacognitive Training for Depression was applied. The adaptation study of the Metacognitive Training for Depression program to Turkish culture was conducted by Okyay and Taş (2017) and the results of the study show that there is a significant difference in the data of Rumi Positive & Negative Scales, Ruminative Reactions Scale and Self-Efficacy Scale in depression patients who were administered this program. In another study (2022), after Metacognitive Training for Depression, there was a decrease in the Beck Depression Scale and Cognitive Distortions Scale scores, depression and cognitive distortion levels of patients.

The presentation of the positive effects of Metacognitive Training for Depression with high level of evidence has contributed to the development of the Metacognitive Training for Older Adults (MCT-Silver) program for depression in older adults. Metacognitive Training-Silver focuses on helping individuals move away from thought patterns that feed/support depression and focuses on physical changes that occur during the aging process, coping with loss and adapting to new social roles. Metacognitive Training-Silver addresses how to identify and reinterpret values in life for individuals aged 60 and over and how to move towards accepting situations that cannot be prevented/changed. In the first pilot study (2018) of the Metacognitive Training-Silver program, a significant reduction in depressive symptoms and dysfunctional attitudes was found. Therefore, more studies are needed to prove the effectiveness of the Metacognitive Training-Silver program.

The Metacognitive Training-Silver program has not yet been adapted to Turkish culture and studies are needed to prove its effectiveness in Turkey. In this direction, a randomized controlled trial is planned to evaluate the effectiveness of the Metacognitive Training-Silver program in older adults diagnosed with depression.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years and over,
* Diagnosis of depression by a psychiatrist according to DSM-V criteria,
* No change in psychopharmacological medications used within 3 months before the Metacognitive Training-Silver program,
* No psychiatric hospitalization in the last 3 months,
* No problems with vision, hearing, and understanding,
* Being literate,

Exclusion Criteria:

* Individuals under 60 years of age,
* Comorbid with a diagnosis of depression to the extent that it interferes with the understanding of the Metacognitive Training-Silver program;

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Beck's Depression Inventory (BDI): Time 1 | BDI will be applied on the first day of Metacognitive Training-Silver to both groups.
  The purpose of the inventory, developed by Aaron T. Beck et al. in 1978, is to measure the severity and change of depressive symptoms in the individual. The Turkish validity and reliability study was carried out by Hisli Şahin. The scale provides a 4-point Likert-type measurement consisting of 21 items. In the scale, the individual is asked to indicate how he or she has felt in the last week. The high score obtained from the scale shows a high level of depression. (Hisli 1989a; Hisli 1989b). The BDI will be used at the beginning of the Metacognitive Training-Silver.
Beck's Depression Inventory (BDI): Time 2 | BDI will be applied after the 8 sessions of Metacognitive Training-Silver completed to both groups. The training will be completed in 8 weeks.
  The purpose of the inventory, developed by Aaron T. Beck et al. in 1978, is to measure the severity and change of depressive symptoms in the individual. The Turkish validity and reliability study was carried out by Hisli Şahin. The scale provides a 4-point Likert-type measurement consisting of 21 items. In the scale, the individual is asked to indicate how he or she has felt in the last week. The high score obtained from the scale shows a high level of depression. (Hisli 1989a; Hisli 1989b). The BDI will be used at the end of the Metacognitive Training-Silver.
Beck's Depression Inventory (BDI): Time 3 | BDI will be reapplied for a follow up evaluation, up to 3 months after the final program, in both groups.
  The purpose of the inventory, developed by Aaron T. Beck et al. in 1978, is to measure the severity and change of depressive symptoms in the individual. The Turkish validity and reliability study was carried out by Hisli Şahin. The scale provides a 4-point Likert-type measurement consisting of 21 items. In the scale, the individual is asked to indicate how he or she has felt in the last week. The high score obtained from the scale shows a high level of depression. (Hisli 1989a; Hisli 1989b). The BDI will be used for follow-up evaluation up to 3 months after the final program.
Dysfunctional Attitude Scale (Revised and Abbreviated Turkish Version- DAS-R-TR): Time 1 | DAS-R-TR will be applied on the first day of Metacognitive Training-Silver to both groups.
  It was developed by Weissman and Beck (1987) as A and B forms, each consisting of 40 items, in order to detect intermediate beliefs that cause depression or anxiety in individuals and to learn their frequency (Weissman and Beck, 1978). However, the validity and reliability study of the revised and abbreviated version of the form was conducted by Batmaz and Özdel (2016) in order to be more useful for practitioners and those who filled out the scale. The scale, which consists of 13 items in the 7-Likert type, has two sub-dimensions as "Perfectionism/Achievement" (first 8 items) and "Need for Approval/Dependency" (last 5 items). If the total scores obtained are high, it indicates that individuals have more dysfunctional attitudes (Batmaz and Özdel, 2016). The DAS-R-TR will be used at the beginning of the Metacognitive Training-Silver.
Dysfunctional Attitude Scale (Revised and Abbreviated Turkish Version- DAS-R-TR): Time 2 | DAS-R-TR will be applied after the 8 sessions of Metacognitive Training-Silver completed to both groups. The training will be completed in 8 weeks.
  It was developed by Weissman and Beck (1987) as A and B forms, each consisting of 40 items, in order to detect intermediate beliefs that cause depression or anxiety in individuals and to learn their frequency (Weissman and Beck, 1978). However, the validity and reliability study of the revised and abbreviated version of the form was conducted by Batmaz and Özdel (2016) in order to be more useful for practitioners and those who filled out the scale. The scale, which consists of 13 items in the 7-Likert type, has two sub-dimensions as "Perfectionism/Achievement" (first 8 items) and "Need for Approval/Dependency" (last 5 items). If the total scores obtained are high, it indicates that individuals have more dysfunctional attitudes (Batmaz and Özdel, 2016). The DAS-R-TR will be used at the end of the Metacognitive Training-Silver.
Dysfunctional Attitude Scale (Revised and Abbreviated Turkish Version- DAS-R-TR): Time 3 | DAS-R-TR will be reapplied for a follow up evaluation, up to 3 months after the final program, in both groups.
  It was developed by Weissman and Beck (1987) as A and B forms, each consisting of 40 items, in order to detect intermediate beliefs that cause depression or anxiety in individuals and to learn their frequency (Weissman and Beck, 1978). However, the validity and reliability study of the revised and abbreviated version of the form was conducted by Batmaz and Özdel (2016) in order to be more useful for practitioners and those who filled out the scale. The scale, which consists of 13 items in the 7-Likert type, has two sub-dimensions as "Perfectionism/Achievement" (first 8 items) and "Need for Approval/Dependency" (last 5 items). If the total scores obtained are high, it indicates that individuals have more dysfunctional attitudes (Batmaz and Özdel, 2016). The DAS-R-TR will be used for follow-up evaluation up to 3 months after the final program.
Metacognition Questionnaire-30 (MCQ-30): Time 1 | MCQ-30 will be applied on the first day of Metacognitive Training-Silver to both groups.
  The MCQ-30 assesses individual differences in unhelpful metacognitions which may contribute to obsessive and compulsive symptoms, pathological worry, and underpin trait anxiety. The scale was developed based on the metacognitive model by Cartwright-Hatton & Wells (65 items, 1997) and was shortened by Wells & Cartwright-Hatton (30 items, 2004). The Turkish study was carried out by Yılmaz et al. and Tosun & Irak in 2008 (Yılmaz et al., 2008; Tosun and Irak, 2008). According to the study of Tosun & Irak (2008), a 4-point Likert-type scale consists five sub-dimensions: (Lack of) Cognitive Confidence, Positive Beliefs about Worry, Cognitive Self-Consciousness, Negative Beliefs about Uncontrollability and Danger, and Need to Control Thoughts. An increase in the score indicates an increase in pathological metacognitive activity (Tosun & Irak, 2008). The MCQ-30 will be used at the beginning of the Metacognitive Training-Silver.
Metacognition Questionnaire-30 (MCQ-30): Time 2 | MCQ-30 will be applied after the 8 sessions of Metacognitive Training-Silver completed to both groups. The training will be completed in 8 weeks.
  The MCQ-30 assesses individual differences in unhelpful metacognitions which may contribute to obsessive and compulsive symptoms, pathological worry, and underpin trait anxiety. The scale was developed based on the metacognitive model by Cartwright-Hatton & Wells (65 items, 1997) and was shortened by Wells & Cartwright-Hatton (30 items, 2004). The Turkish study was carried out by Yılmaz et al. and Tosun & Irak in 2008 (Yılmaz et al., 2008; Tosun and Irak, 2008). According to the study of Tosun & Irak (2008), a 4-point Likert-type scale consists five sub-dimensions: (Lack of) Cognitive Confidence, Positive Beliefs about Worry, Cognitive Self-Consciousness, Negative Beliefs about Uncontrollability and Danger, and Need to Control Thoughts. An increase in the score indicates an increase in pathological metacognitive activity (Tosun & Irak, 2008). The MCQ-30 will be used at the end of the Metacognitive Training-Silver.
Metacognition Questionnaire-30 (MCQ-30): Time 3 | MCQ-30 will be applied on the first day of Metacognitive Training-Silver to both groups.
  The MCQ-30 assesses individual differences in unhelpful metacognitions which may contribute to obsessive and compulsive symptoms, pathological worry, and underpin trait anxiety. The scale was developed based on the metacognitive model by Cartwright-Hatton & Wells (65 items, 1997) and was shortened by Wells & Cartwright-Hatton (30 items, 2004). The Turkish study was carried out by Yılmaz et al. and Tosun & Irak in 2008 (Yılmaz et al., 2008; Tosun and Irak, 2008). According to the study of Tosun & Irak (2008), a 4-point Likert-type scale consists five sub-dimensions: (Lack of) Cognitive Confidence, Positive Beliefs about Worry, Cognitive Self-Consciousness, Negative Beliefs about Uncontrollability and Danger, and Need to Control Thoughts. An increase in the score indicates an increase in pathological metacognitive activity (Tosun & Irak, 2008). The MCQ-30 will be used for follow-up evaluation up to 3 months after the final program.
The WHO-Europe Attitudes of Aging Questionnaire (EAAQ): Time 1 | EAAQ will be applied on the first day of Metacognitive Training-Silver to both groups.
  The attitudes to ageing questionnaire was developed to provide a standard way of measuring attitudes to ageing from the perspective of older people. The scale was developed within the scope of a multi-center project supported by the EU 5th Framework Program to determine the perception level to aging of elderly. The Turkish adaptation and psychometric properties of the scale were studied by Eser et al. in 2011. The scale is a 5-point Likert-type scale consisting of three sub-dimensions (Psychosocial Loss; Physical Change and Psychological Growth) and a total of 24 items. As the total score of the scale increases, the attitude towards the related dimension also increases positively. (Eser et al. 2011). The EAAQ will be used at the beginning of the Metacognitive Training-Silver.
The WHO-Europe Attitudes of Aging Questionnaire (EAAQ): Time 2 | EAAQ will be applied after the 8 sessions of Metacognitive Training-Silver completed to both groups. The training will be completed in 8 weeks.
  The attitudes to ageing questionnaire was developed to provide a standard way of measuring attitudes to ageing from the perspective of older people. The scale was developed within the scope of a multi-center project supported by the EU 5th Framework Program to determine the perception level to aging of elderly. The Turkish adaptation and psychometric properties of the scale were studied by Eser et al. in 2011. The scale is a 5-point Likert-type scale consisting of three sub-dimensions (Psychosocial Loss; Physical Change and Psychological Growth) and a total of 24 items. As the total score of the scale increases, the attitude towards the related dimension also increases positively. (Eser et al. 2011). The EAAQ will be used at the end of the Metacognitive Training-Silver.
The WHO-Europe Attitudes of Aging Questionnaire (EAAQ): Time 3 | EAAQ will be applied on the first day of Metacognitive Training-Silver to both groups.
  The attitudes to ageing questionnaire was developed to provide a standard way of measuring attitudes to ageing from the perspective of older people. The scale was developed within the scope of a multi-center project supported by the EU 5th Framework Program to determine the perception level to aging of elderly. The Turkish adaptation and psychometric properties of the scale were studied by Eser et al. in 2011. The scale is a 5-point Likert-type scale consisting of three sub-dimensions (Psychosocial Loss; Physical Change and Psychological Growth) and a total of 24 items. As the total score of the scale increases, the attitude towards the related dimension also increases positively. (Eser et al. 2011). The EAAQ will be used for follow-up evaluation up to 3 months after the final program.

SECONDARY OUTCOMES:
Personal Information Form (Sociodemographic Characteristics and Clinical Data) | Personal Information Form will be applied on the first day of the first session of Metacognitive Training-Silver on both groups.
  The personal information form prepared by the researchers is a 16-question form containing sociodemographic characteristics such as age, gender, marital status, educational status, and depression-related clinical data such as diagnosis time, and treatment method (pharmacotherapy and/or psychotherapy) etc. This form will be applied on the first day of the program to all participants and will be collected once.

CONTACTS AND LOCATIONS:
Overall Officials: Merve MURAT MEHMED ALİ, MSc, RN, Principal Investigator — Istanbul University - Cerrahpasa; Sevim BUZLU, Prof, PhD, RN, Study Chair — Istanbul University - Cerrahpasa; Lara Guedes de Pinho, Assoc Prof, PhD, RN, Study Chair — University of Évora
Locations (1):
- Istanbul University - Cerrahpaşa, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD (Individual Participant Data) available. After the study is completed, the publication which includes the data results will be available.

REFERENCES:
- [Background] Batmaz S, Ozdel K. Psychometric Properties of the Revised and Abbreviated form of the Turkish Version of the Dysfunctional Attitude Scale. Psychol Rep. 2016 Feb;118(1):180-198. doi: 10.1177/0033294116628349. PMID 29693528
- [Background] COVID-19 Mental Disorders Collaborators. Global prevalence and burden of depressive and anxiety disorders in 204 countries and territories in 2020 due to the COVID-19 pandemic. Lancet. 2021 Nov 6;398(10312):1700-1712. doi: 10.1016/S0140-6736(21)02143-7. Epub 2021 Oct 8. PMID 34634250
- [Background] Cuijpers P, Sijbrandij M, Koole SL, Andersson G, Beekman AT, Reynolds CF 3rd. Adding psychotherapy to antidepressant medication in depression and anxiety disorders: a meta-analysis. World Psychiatry. 2014 Feb;13(1):56-67. doi: 10.1002/wps.20089. PMID 24497254
- [Background] Evans-Lacko S, Aguilar-Gaxiola S, Al-Hamzawi A, Alonso J, Benjet C, Bruffaerts R, Chiu WT, Florescu S, de Girolamo G, Gureje O, Haro JM, He Y, Hu C, Karam EG, Kawakami N, Lee S, Lund C, Kovess-Masfety V, Levinson D, Navarro-Mateu F, Pennell BE, Sampson NA, Scott KM, Tachimori H, Ten Have M, Viana MC, Williams DR, Wojtyniak BJ, Zarkov Z, Kessler RC, Chatterji S, Thornicroft G. Socio-economic variations in the mental health treatment gap for people with anxiety, mood, and substance use disorders: results from the WHO World Mental Health (WMH) surveys. Psychol Med. 2018 Jul;48(9):1560-1571. doi: 10.1017/S0033291717003336. Epub 2017 Nov 27. PMID 29173244
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Background] Hu T, Zhao X, Wu M, Li Z, Luo L, Yang C, Yang F. Prevalence of depression in older adults: A systematic review and meta-analysis. Psychiatry Res. 2022 May;311:114511. doi: 10.1016/j.psychres.2022.114511. Epub 2022 Mar 16. PMID 35316691
- [Background] Islam N, Sharp SJ, Chowell G, Shabnam S, Kawachi I, Lacey B, Massaro JM, D'Agostino RB Sr, White M. Physical distancing interventions and incidence of coronavirus disease 2019: natural experiment in 149 countries. BMJ. 2020 Jul 15;370:m2743. doi: 10.1136/bmj.m2743. PMID 32669358
- [Background] Jelinek L, Hauschildt M, Wittekind CE, Schneider BC, Kriston L, Moritz S. Efficacy of Metacognitive Training for Depression: A Randomized Controlled Trial. Psychother Psychosom. 2016;85(4):231-4. doi: 10.1159/000443699. Epub 2016 May 27. No abstract available. PMID 27230865
- [Background] Jelinek L, Van Quaquebeke N, Moritz S. Cognitive and Metacognitive Mechanisms of Change in Metacognitive Training for Depression. Sci Rep. 2017 Jun 14;7(1):3449. doi: 10.1038/s41598-017-03626-8. PMID 28615651
- [Background] Jelinek L, Faissner M, Moritz S, Kriston L. Long-term efficacy of Metacognitive Training for Depression (D-MCT): A randomized controlled trial. Br J Clin Psychol. 2019 Sep;58(3):245-259. doi: 10.1111/bjc.12213. Epub 2018 Dec 16. PMID 30556583
- [Background] Liu YC, Tang CC, Hung TT, Tsai PC, Lin MF. The Efficacy of Metacognitive Training for Delusions in Patients With Schizophrenia: A Meta-Analysis of Randomized Controlled Trials Informs Evidence-Based Practice. Worldviews Evid Based Nurs. 2018 Apr;15(2):130-139. doi: 10.1111/wvn.12282. Epub 2018 Feb 28. PMID 29489070
- [Background] Moritz S, Woodward TS. Metacognitive training in schizophrenia: from basic research to knowledge translation and intervention. Curr Opin Psychiatry. 2007 Nov;20(6):619-25. doi: 10.1097/YCO.0b013e3282f0b8ed. PMID 17921766
- [Background] Perini G, Cotta Ramusino M, Sinforiani E, Bernini S, Petrachi R, Costa A. Cognitive impairment in depression: recent advances and novel treatments. Neuropsychiatr Dis Treat. 2019 May 10;15:1249-1258. doi: 10.2147/NDT.S199746. eCollection 2019. PMID 31190831
- [Background] Skoog I. COVID-19 and mental health among older people in Sweden. Int Psychogeriatr. 2020 Oct;32(10):1173-1175. doi: 10.1017/S104161022000143X. Epub 2020 Jul 8. No abstract available. PMID 32635950
- [Background] van Oosterhout B, Smit F, Krabbendam L, Castelein S, Staring AB, van der Gaag M. Metacognitive training for schizophrenia spectrum patients: a meta-analysis on outcome studies. Psychol Med. 2016 Jan;46(1):47-57. doi: 10.1017/S0033291715001105. Epub 2015 Jul 20. PMID 26190517
- [Background] Yilmaz AE, Gencoz T, Wells A. Psychometric characteristics of the Penn State Worry Questionnaire and Metacognitions Questionnaire-30 and metacognitive predictors of worry and obsessive-compulsive symptoms in a Turkish sample. Clin Psychol Psychother. 2008 Nov-Dec;15(6):424-39. doi: 10.1002/cpp.589. PMID 19115461
- [Background] Dietrichkeit M, Moritz S, Jelinek L. Die Behandlung psychischer Störungen mittels metakognitiver Interventionen am Beispiel des Metakognitiven Trainings für Depression (D-MKT). [The treatment of mental disorders using metacognitive interventions using the example of Metacognitive Training for Depression (D-MKT)]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie. 2020; 68: 160-170.
- [Background] Erdfelder E, Faul F, Buchner A. GPOWER: A general power analysis program. Behavior Research Methods, Instruments & Computers. 1996; 28(1): 1-11.
- [Background] Eser E, Gerçeklioğlu Saatli G, Eser S, Fidaner C, Baysan P, Pala T, Dündar P. Dünya sağlık örgütü - Avrupa "yaşlanma tutumu anketi (AAQ)" Türkçe sürümünün (AYTA-TR) psikometrik özellikleri. Türk Geriatri Dergisi. 2011; 14(2): 101 - 110.
- [Background] Falci SG, Marques LS. CONSORT: when and how to use it. Dental Press J Orthod. 2015 May-Jun;20(3):13-5. doi: 10.1590/2176-9451.20.3.013-015.ebo. No abstract available. PMID 26154451
- [Background] Fansi A, Jehanno C, Lapalme M, Drapeau M, Bouchard S. [Effectiveness of psychotherapy compared to pharmacotherapy for the treatment of anxiety and depressive disorders in adults: A literature review]. Sante Ment Que. 2015 Winter;40(4):141-73. French. PMID 27203537
- [Background] Hisli N. Beck Depresyon Envanterinin Üniversite Öğrencileri İçin Geçerliği Güvenirliği, Psikoloji Dergisi. 1989; 23: 3-13.
- [Background] Hisli N. Beck Depresyon Envanterinin Geçerliği Üzerine Bir Çalışma. Psikoloji Dergisi. 1989; 22: 118-126.
- [Background] Jelinek L, Otte C, Arlt S, Hauschildt M. Denkverzerrungen erkennen und korrigieren: Eine Machbarkeitsstudie zum Metakognitiven Training bei Depressionen (D-MKT). [Identifying and correcting cognitive biases: a pilot study on the Metacognitive Training for Depression (D-MCT)]. Zeitschrift für Psychiatrie, Psychologie und Psychotherapie. 2013; 61: 1-8.
- [Background] Kamber O. Depresyon tedavisinde metakognisyon eğitimi grup terapisinin (D-MKT) Türk Kültüründeki etkinliği [master's thesis]. [İstanbul (TR)]: Üsküdar Üniversitesi; 2017.
- [Background] Özgüç S, Tanriverdi D. Effects of Metacognitive Training (D-MCT) on Metacognition and Ruminative Thought Levels of Major Depression Patients. Int J Ment Health Addiction. 2023; 21, 2017-2028.
- [Background] Schneider BC, Bücker L, Riker S, Jelinek L. A pilot study of Metacognitive Training for Depression in older adults. Zeitschrift für Neuropsychologie. 2018; 29: 7-19.
- [Background] Tosun A, Irak M. [Adaptation, validity, and reliability of the Metacognition Questionnaire-30 for the Turkish population, and its relationship to anxiety and obsessive-compulsive symptoms]. Turk Psikiyatri Derg. 2008 Spring;19(1):67-80. Turkish. PMID 18330745
- [Background] Jelinek L, Hauschildt M, Moritz S. Metakognitives Training bei Depression. Weinheim: Beltz; 2015.
- [Background] Amerikan Psikiyatri Birliği, 2015. Ruhsal bozuklukların tanısal ve sayımsal el kitabı (E. Köroğlu.). Hekimler Yayın Birliği, 2013. ISBN-10: 9753001983, ISBN-13: 978-9753001984
- See also: Institute of Health Metrics and Evaluation, 2022, Global health data exchange results — http://ghdx.healthdata.org/gbd-results-tool?params=gbd-api-2019-permalink/d780dffbe8a381b25e1416884959e88b
- See also: World Health Organization, 2022, World Health Statistics 2022 — https://www.who.int/news/item/20-05-2022-world-health-statistics-2022
- See also: World Health Organization, 2021, Depression — https://www.who.int/news-room/fact-sheets/detail/depression